CLINICAL TRIAL: NCT03202719
Title: Duration of Priming and Antibody Decay With Full-dose Inactivated Poliovirus Vaccine (IPV) Administered With or Without Bivalent Oral Poliovirus Vaccine (bOPV)
Brief Title: Duration of IPV Priming and Antibody Decay
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ICDDRB-RRC-PR-17034
Record Dates: First submitted 2017-06-23; First posted 2017-06-29 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Poliomyelitis
Keywords: Inactivated polio vaccine; Polio; oral polio vaccine
MeSH Terms: conditions — Poliomyelitis | interventions — Aging; Poliovirus Vaccine, Inactivated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- IPV at ages 14 weeks and 18 months (Active Comparator): Participants in this arm will receive bivalent oral poliovirus vaccine (bOPV) at 6, 10 and 14 weeks of age and inactivated poliovirus vaccine (IPV) at 14 weeks and 18 months of age
  Interventions: Biological: Bivalent oral poliovirus vaccine (bOPV) at 6,10 and 14 weeks of age; Biological: Inactivated poliovirus vaccine (IPV) at 14 weeks and 18 months of age
- IPV at ages 14 weeks, 18 weeks and 18 months (Active Comparator): Participants in this arm will receive bivalent oral poliovirus vaccine (bOPV) at 6, 10 and 14 weeks of age and inactivated poliovirus vaccine (IPV) at 14 weeks, 18 weeks and 18 months of age
  Interventions: Biological: Bivalent oral poliovirus vaccine (bOPV) at 6,10 and 14 weeks of age; Biological: Inactivated poliovirus vaccine (IPV) at 14 weeks, 18 weeks and 18 months of age
- IPV at ages 14 weeks and 9 months (Active Comparator): Participants in this arm will inactivated poliovirus vaccine (IPV) at 14 weeks and 9 months of age
  Interventions: Biological: Inactivated poliovirus vaccine (IPV) at 14 weeks and 9 months of age
- IPV at ages 6 weeks and 9 months (Active Comparator): Participants in this arm will inactivated poliovirus vaccine (IPV) at 6 weeks and 9 months of age
  Interventions: Biological: Inactivated poliovirus vaccine (IPV) at 6 weeks and 9 months of age
- IPV at ages 6 and 14 weeks (Active Comparator): Participants in this arm will inactivated poliovirus vaccine (IPV) at 6 and 14 weeks of age
  Interventions: Biological: Inactivated poliovirus vaccine (IPV) at 6 and 14 weeks of age

INTERVENTIONS:
Biological: Bivalent oral poliovirus vaccine (bOPV) at 6,10 and 14 weeks of age — bOPV at 6, 10 and 14 weeks of age
  Arms: IPV at ages 14 weeks and 18 months; IPV at ages 14 weeks, 18 weeks and 18 months
Biological: Inactivated poliovirus vaccine (IPV) at 14 weeks and 18 months of age — IPV at 14 weeks and 18 months of age
  Arms: IPV at ages 14 weeks and 18 months
Biological: Inactivated poliovirus vaccine (IPV) at 14 weeks, 18 weeks and 18 months of age — IPV at 14 weeks, 18 weeks and 18 months of age
  Arms: IPV at ages 14 weeks, 18 weeks and 18 months
Biological: Inactivated poliovirus vaccine (IPV) at 14 weeks and 9 months of age — IPV at 14 weeks and 9 months of age
  Arms: IPV at ages 14 weeks and 9 months
Biological: Inactivated poliovirus vaccine (IPV) at 6 weeks and 9 months of age — IPV at 6 weeks and 9 months of age
  Arms: IPV at ages 6 weeks and 9 months
Biological: Inactivated poliovirus vaccine (IPV) at 6 and 14 weeks of age — IPV at 6 and 14 weeks of age
  Arms: IPV at ages 6 and 14 weeks

SUMMARY:
This is an open-label randomized phase IV clinical trial assessing immunogenicity of poliovirus vaccines.Participants will be enrolled at 6 weeks of age and followed to 18 months of age. The study will recruit 1645 participants in five arms.

DETAILED DESCRIPTION:
Poliomyelitis is an acute infection caused by polioviruses. Oral poliovirus vaccines are live attenuated viral vaccines and the vaccine virus in OPV can mutate and acquire neurovirulence causing paralysis either due to vaccine-associated paralytic polio (VAPP) or due to circulating vaccine-derived polioviruses (cVDPV), in which the attenuated vaccine virus not only acquires the ability to cause paralysis but can also circulate similar to wild poliovirus (WPV). Therefore, polio eradication will require eventual cessation of all OPVs.

Wild poliovirus type 2 (WPV2) was declared eradicated in September 2015. Since then paralysis associated with type 2 poliovirus has continued mainly due to vaccine derived polio viruses (VDPVs) from type 2 OPV (OPV2). Due to the continued threat of paralysis from a mutated, neurovirulent and vaccine-derived type 2 poliovirus, the Strategic Advisory Group of Experts on Immunization (SAGE), a global advisory committee on immunization, recommended a phased cessation of OPV starting with OPV2. By May 2016, OPV2 was successfully withdrawn globally when trivalent OPV (tOPV) was replaced with bivalent OPV (bOPV), which was preceded by a phased introduction of inactivated poliovirus vaccine (IPV). SAGE has recommended at least one dose of IPV at age ≥14 weeks because IPV immunogenicity is expected to be highest after maternal antibodies have declined by age 14 weeks. However, studies have not assessed if priming after one IPV dose declines over time.

Types 1 and 3 OPV cessation is likely expected in 2020-2022, i.e. 1-2 years after certification of global interruption of wild poliovirus transmission. After cessation of bOPV, IPV will be used for routine polio vaccination for 5-10 years.Recently, SAGE recommended that IPV be used after global OPV withdrawal with an IPV schedule that achieves at least 90% seroconversion with two full or fractional doses. SAGE has recommended that the first dose be administered after 14 weeks of age and an interval of at least 4 months between two IPV doses. In the proposed clinical trial, immunogenicity of two IPV doses with schedules that are likely to achieve 90% immune response to all poliovirus types is being assessed to inform SAGE policy deliberations on potential IPV schedules after OPV cessation. A head-to-head comparison of different IPV schedules is important to determine the immunogenicity of the schedules under similar conditions and evaluate the differences in population immunity, a product of immunogenicity and vaccination coverage, with the different IPV schedules.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants 6 weeks of age (range: 42-48 days).
* Parents that consent for participation in the full length of the study.
* Parents that are able to understand and comply with planned study procedures.

Exclusion Criteria:

* Parents and infants who are unable to participate in the full length of the study.
* A diagnosis or suspicion of immunodeficiency disorder either in the infant or in an immediate family member.
* A diagnosis or suspicion of bleeding disorder that would contraindicate parenteral administration of IPV or collection of blood by venipuncture.
* Acute diarrhoea, infection or illness at the time of enrollment (6 weeks of age) that would require infant's admission to a hospital.
* Acute vomiting and intolerance to liquids within 24 hours before the enrollment visit (6 weeks of age).
* Evidence of a chronic medical condition identified by a study medical officer during physical exam.
* Receipt of any polio vaccine (OPV or IPV) before enrollment based upon documentation or parental recall.
* Known allergy/sensitivity or reaction to polio vaccine, or its contents.
* Infants from multiple births. Infants from multiple births will be excluded because the infant(s) who is/are not enrolled would likely receive OPV through routine immunization and transmit vaccine poliovirus to the enrolled infant.
* Infants from premature births (<37 weeks of gestation).

Ages: 6 Weeks to 7 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1645 (Actual)
Dates: Start 2017-11-05 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Immunogenicity of IPV vaccination schedule | Change after receiving vaccine compared to that at 6 weeks of age
  Immunogenicity will be assessed by measuring type-specific poliovirus antibody titers and assessing the change in antibody titers after receiving study vaccine compared to 6 weeks of age. The cumulative proportion of participants who demonstrate an immune response one month after receiving the last IPV dose of the experimental schedule. Immune response will be defined as either seronegative participants (<1:8 titers) who become seropositive (≥1:8) [seroconversion] or participants who demonstrate a four-fold increase in titer (boosting).
Poliovirus type 2 priming with IPV | Proportion who demonstrate type 2 response at 18 months and 1 week among those who did not respond at 19 weeks
  The proportion of participants who demonstrate type 2 immune response one week after receiving an additional IPV dose (secondary vaccination) after the proposed primary IPV vaccination series will be determined. Priming is the proportion of participants that demonstrate type 2 immune response among those who have not previously responded to the primary IPV vaccination series.

CONTACTS AND LOCATIONS:
Locations (2):
- Bangladesh (2):
  - International Center for Diarrhoeal Disease Research, Bangladesh, Dhaka
  - Mirpur clinic (International Center for Diarrhoeal Disease Research, Bangladesh), Dhaka

IPD SHARING:
Plan to Share IPD: No
Summary tables to be shared December 2019